CLINICAL TRIAL: NCT05530811
Title: Comparative Study Between Dexamethasone Plus Bupivacaine Versus Bupivacaine in Management of Suprazygomatic Maxillary Nerve Block in Cleft Palate Patients.
Brief Title: Dexamethasone as Adjuvant to Bupivacaine in Suprazygomatic Maxillary Nerve Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mark Wageh, Anaesthesia and ICU Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: suprazygomatic maxillary nerve
Record Dates: First submitted 2021-11-17; First posted 2022-09-07 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Nerve Block
MeSH Terms: interventions — Dexamethasone; Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with dexamethasone (Active Comparator): bilateral suprazygomatic maxillary nerve block will be performed with 1 mL of 0.5% bupivacaine was added to 0.1 mg.kg-1 dexamethasone and diluted to 2 mL with 0.9% saline.
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine
- without dexamethasone (Placebo Comparator): bilateral suprazygomatic maxillary nerve block will be performed with 1 mL of 0.5% bupivacaine alone and diluted to 2 mL with 0.9% saline.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexamethasone — The suprazygomatic maxillary nerve block approach will be performed with a 27-gauge 38-mm needle following aseptic preparation of the skin and using the anatomical landmarks. The puncture site will be at the frontozygomatic angle formed by the zygomatic arch and posterior orbital rim. After inserting the needle perpendicular to the skin and contacting the greater wing of the sphenoid (approximately 20 mm deep), the needle will be partially withdrawn, reoriented approximately 20° anterior and 10° inferior, and advanced 35 to 38 mm to direct the needle into the pterygopalatine fossa. After negative blood aspiration, the prepared solution will be injected over 20 s on each side. Massage of injection point with pressure for 2 min will be done. No additional local anesthetic will be injected by the surgeon either peri-incisional or submucosal.
  Arms: with dexamethasone
Drug: Bupivacaine — 0.5% bupivacaine

SUMMARY:
Postoperative pain score, Faces, Legs, Activity, Cry, Consolability (FLACC) is the primary outcome. The secondary outcomes are the first-time requested analgesia, the number of children required analgesia, the total amount of analgesic requirements during first the 24 hours.

DETAILED DESCRIPTION:
Congenital cleft palate (CP) occurs in children at a rate of about 1.5 per 10 000 births , requiring early surgery, during the first months of life. The surgical procedure can be complicated by airway obstruction and respiratory complications. CP is painful in the first 24-48 hours following surgery.

Different treatment modalities have been used for reducing or ameliorating the pain following cleft palate repair. These include opioids, paracetamol, non steroidal anti-inflammatory drugs (NSAIDs). However, the analgesic drugs may provide inadequate analgesia and have side effects such as respiratory depression and bleeding. The inherent disadvantages of analgesic pharmacotherapy in children promoted interest in nerve blocking techniques for operative analgesia.

The maxillary nerve, the second division of the trigeminal nerve, leaves the cranial part of the face through the foramen rotundum, and then passes forward and laterally through the pterygopalatine fossa, at the bottom of the pterygomaxillary fossa, and reaches the floor of the orbit by the infra-orbital foramen. This sensory nerve supplies innervation of the lower eyelid, the upper lip, the skin between them, the roof of the mouth, and the palate. Bilateral infra-orbital nerve block is clearly inefficient for anesthesia of the posterior part of the palate (hard palate). The infrazygomatic route of the maxillary block, useful for trigeminal neuralgia, can present several risks such as penetration of the orbit or the skull and accidental maxillary artery puncture. The palatine nerve block could be efficient for analgesia following cleft palate repair, but the technique requires identifying the first molar, which is absent in infants. Finally, submucosal infiltration performed by the surgeon seems to alter surgical conditions. Maxillary nerve block using the suprazygomatic approach has demonstrated beneficial effects in adults for trigeminal neuralgia and limits the risks related to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 and 9 years
* Children scheduled for primary surgery for soft palate cleft or soft and hard palate clefts
* Gender: both
* ASA grade I - II.
* Informed consent.

Exclusion Criteria:

* Parent refusal
* History of developmental delay or mental retardation, which will make observational pain intensity assessment difficult
* Hypersensitivity to any local anesthetics
* Bleeding diathesis
* Children with co-morbid conditions like congenital heart disease, respiratory pathology and central nervous system disorders
* Skin lesions or wounds at the puncture site of the proposed block

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score | baseline
  pain in Faces, Legs, Activity, Cry, Consolability (FLACC) Each category is scored on the 0-2 scale which results in a total score of 0-10.
Assessment of Behavioral Score | baseline
  0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain

SECONDARY OUTCOMES:
The first-time requested analgesia . | 24 hours
  The first-time requested analgesia .
The number of children required analgesia. | 24 hours
  The number of children required analgesia.
The total amount of analgesic requirements . | 24 hours
  The total amount of analgesic requirements .